CLINICAL TRIAL: NCT04831112
Title: A Comparative Study Between the Use of Topical Honey and EUSOL Dressing in Necrotizing Fascitis Wounds
Brief Title: Compare Effects of Dressing With Honey and EUSOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Lajpat Rai, Principal Investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-1491/DUHS/Approval/2020
Record Dates: First submitted 2021-03-21; First posted 2021-04-05 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Necrotizing Fascitis; Wound Infection
MeSH Terms: conditions — Fasciitis, Necrotizing; Wound Infection | interventions — Honey; Eusol

STUDY DESIGN:
Intervention Model Description: Experimental randomised trial
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Honey (Experimental): Topical honey to be used for dressing 4ml per square inch.
  Interventions: Drug: Honey; Combination Product: EUSOL
- EUSOL (Active Comparator): EUSOL soaked gauze to be placed over the wound as dressing.
  Interventions: Drug: Honey; Combination Product: EUSOL

INTERVENTIONS:
Drug: Honey — Dressing of necrotizing fascitis wounds with honey.
Combination Product: EUSOL — Dressing of necrotizing fascitis wounds with EUSOL.

SUMMARY:
Honey is super saturated solution containing sugar derived from nectar gathered by honeybee. Honey is viscus supersaturated solution mainly composed of sugar and water along with minor constituents such as minerals, vitamins, amino acids, organic acids, flavonoids, and other phenolic compound and aromatic substances. Honey contents according to percentages are fructose 38.6%, glucose 31%, water 17%, lactose 7.2%, larger sugars 4.7% and rest of micronutrients and elemental compounds are 1.5%. Honey enhances wound healing by removing slough and necrotic tissue from wound. It promotes wound healing by increasing angiogenesis, granulation and epithelization. Honey possess antimicrobial activity against bacteria like methicillin resistant staphylococcus aureus, vancomycin resistant Escherichia Coli, pseudomonas aeruginosa, and many other species. It also has activity against some yeast species such as aspergillus and penicillium.

Honey used for dressing will be 'Langnese Honey". Langnese honey is raw honey / unprocessed packed as collected, quality and quantity will be same for patients.

DETAILED DESCRIPTION:
This prospective randomized trial will be conducted in all patients undergoing dressing after debridement of necrotizing fasciitis wounds. Study will be conducted for 6 months after approval IRB. Patient will be inducted through emergency department. After debridement, patient will be enrolled in study via simple random sampling for dressing with either EUSOL or Honey. Honey quantity for wound will be 4ml per square inch. In patient whose both limbs involved by necrotizing fasciitis, after debridement, dressing will be done with honey in one limb and EUSOL in other limb. Patient will be enrolled in study whose debridement already done.

EUSOL is solution commonly used for dressing of wounds. Honey is also used for dressing of wounds. Honey is a viscous, supersaturated sugar derived from nectar gathered by a honeybee. Honey enhances wound healing by providing moist environment, antibacterial activity, deodorizes, decrease inflammation, edema and exudation. Honey increase rate of wound healing by promoting angiogenesis, granulation and epithelization. Dressing will be done by residents of our ward under supervision of faculty. At first time of debridement pus or tissue will be sent for culture and sensitivity meanwhile broad-spectrum antibiotic will be started. Once dressing will started, wide wound span will be measured and assessed daily for granulation tissue and removal of slough. Questionnaire will be filled by PI for allergic reaction to solution, appearance of granulation tissue and hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years and <70 years.
* Necrotizing fasciitis wounds
* Wide span of wound <20cm

Exclusion Criteria:

* Diabetic Foot wounds
* Traumatic wounds

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 326 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Early wound healing | 3 weeks
  Early wound healing is measured via appearance of granulation tissue over the wound.

SECONDARY OUTCOMES:
Decreased hospital stay | 4 weeks
  Decrease of hospital stay is determined via early discharge of patient from hospital and managed as out patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Dr Ruth K.M Pfau Civil Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No